CLINICAL TRIAL: NCT07076199
Title: A 26-week Study Comparing the Efficacy and Safety of Once-weekly Insulin Icodec and Once-daily Insulin Glargine U100, Both in Combination With Insulin Aspart, in Adults With Type 1 Diabetes
Brief Title: A Research Study to See How a Weekly Insulin, Insulin Icodec, Helps in Reducing the Blood Sugar Compared to Daily Insulin Glargine, Both in Combination With Insulin Aspart, in Adults With Type 1 Diabetes
Acronym: ONWARDS 11
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1436-8182; U1111-1310-7017 (Other: World Health Organization (WHO)); 2024-519945-31 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin icodec; Insulin Glargine; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Insulin icodec + insulin aspart (Experimental): Participants will receive subcutaneously once weekly insulin icodec in combination with 2-4 times daily insulin aspart .
  Interventions: Drug: Insulin icodec; Drug: Insulin aspart
- Insulin glargine+ insulin aspart (Active Comparator): Participants will receive subcutaneously once daily insulin glargine in combination with 2-4 times daily insulin aspart.
  Interventions: Drug: Insulin glargine; Drug: Insulin aspart

INTERVENTIONS:
Drug: Insulin icodec — Insulin icodec will be administered as subcutaneous injection
  Arms: Insulin icodec + insulin aspart
Drug: Insulin glargine — Insulin glargine will be administered as subcutaneous injection.
  Arms: Insulin glargine+ insulin aspart
Drug: Insulin aspart — Insulin aspart will be administered as a subcutaneous injection.

SUMMARY:
This study compares insulin icodec, an insulin taken once a week to insulin glargine, an insulin taken once a day. The study medicine will be investigated in participants with type 1 diabetes. The study will look at how well insulin icodec taken weekly controls blood sugar compared to insulin glargine taken daily. The study will last for about 8.5 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 1 diabetes mellitus greater than or equal to (≥) 1 year before screening.
* Treated with multiple daily insulin injections (daily basal insulin analogue and bolus insulin analogue regimen) ≥ 6 months before screening.
* HbA1c from 7.0-10.0 percentage (%) (53.0-85.8 millimoles per mole (mmol/mol)), both inclusive, at screening confirmed by central laboratory analysis.
* Ability and willingness to adhere to the protocol including performance of self-measured plasma glucose (SMPG) profiles, based on the investigator's judgement.

Exclusion Criteria:

* Known or suspected hypersensitivity to study intervention(s) or related products.
* Previous participation in this study. Participation is defined as signed informed consent.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using adequate contraceptive method.
* Exposure to an investigational medicinal product within 90 days or 5 half-lives of the investigational medicinal product (if known), whichever is longer, before screening.
* Any condition, except for conditions associated with type 1 diabetes mellitus, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Anticipated initiation or anticipated change in concomitant medications (for more than 15 consecutive days) known to affect weight or glucose metabolism (e.g., treatment with thyroid hormones, or systemic corticosteroids).
* Known hypoglycaemic unawareness as indicated by the Investigator according to Clarke's questionnaire question.
* Recurrent severe hypoglycaemic episodes within the last year as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 877 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-11-23 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Change in glycosylated haemoglobin (HbA1c) | From baseline (week 0) to week 26
  Measured in percentage (%)-points.

SECONDARY OUTCOMES:
Change in time in range 3.9-10.0 millimoles per liter (mmol/L) (70-180 milligrams per deciliter (mg/dL)) | From baseline (week-2-0) to week 22-26
  Measured in %-points.
Time spent less than (<)3.0 mmol/L (54 mg/dL) | From week 22 to week 26
  Measured in % of time.
Change in time spent greater than (>)10.0 mmol/L (180 mg/dL) | From baseline (week-2-0) to week 22-26
  Measured in %-points.
Number of severe hypoglycaemic episodes (level 3) | From baseline (week 0) to week 31
  Measured as number of episodes.
Number of clinically significant hypoglycaemicepisodes (level 2) (<3.0mmol/L [54 mg/dL],confirmed by blood glucose (BG) meter) | From baseline (week 0) to week 31
  Measured as number of episodes.
Number of clinically significant hypoglycaemic episodes (level 2) (< 3.0 mmol/L [54 mg/dL], severe hypoglycaemic confirmed by BG meter) or episodes (level 3) | From baseline (week 0) to week 31
  Measured as number of episodes.
Number of continuous glucose continuous glucose (CGM)-based clinically significant hypoglycaemic episodes (level 2) (< 3.0 mmol/L [54 mg/dL]) | From baseline (week 0) to week 31
  Measured as number of episodes.
Mean total weekly insulin dose | From week 24 to week 26
  Measured in insulin units.
Change in body weight | From baseline (week 0) to week 26
  Measured in Kilogram (kg).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (176):
- United States (96):
  - Cullman Clinical Trials, Cullman, Alabama
  - John Muir Health, Concord, California
  - Headlands Research California, LLC, Escondido, California
  - Clinical Res of Central Ca, Fresno, California
  - Providence Medical Foundation, Fullerton, California
  - Scripps Whittier Diabetes Inst, La Jolla, California
  - Loma Linda University Faculty Medical Clinics, Loma Linda, California
  - Pacific Clinical Studies, Los Alamitos, California
  - Pasadena Clinical Trials, Pasadena, California
  - WestenU Health, Pomona, California
  - Alliance Clinical Network, San Diego, California
  - Mills Health Center, San Mateo, California
  - Center for Endocrine DM and Metabolic Disorders, Santa Clarita, California
  - University Clin Investigators, Tustin, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Denver Endocrinology Diabetes and Thyroid Center, Englewood, Colorado
  - Optumcare Clinical Trials,LLC-Golden, Golden, Colorado
  - Northeast Research Institute, Fleming Island, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - West Orange Endocrinology, Ocoee, Florida
  - Suncoast Clinical Research, Inc., Palm Harbor, Florida
  - SRA Trials-Broward, Pembroke Pines, Florida
  - Hanson Clinical Research Center, Port Charlotte, Florida
  - Latin Clinical Trial Ctr, Tamarac, Florida
  - Bayside Clinical Research, Tampa, Florida
  - Metabolic Research Institute Inc, West Palm Beach, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Centricity Research Columbus, Columbus, Georgia
  - Physicians Research Assoc. LLC, Lawrenceville, Georgia
  - Endocrine Research Solutions, Inc, Roswell, Georgia
  - Rocky Mt Clin Res, LLC, Idaho Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - University Of Chicago, Chicago, Illinois
  - Endeavor Health, Skokie, Illinois
  - Indiana Uni School of Med-Ped, Indianapolis, Indiana
  - Iowa Diabetes Research, Des Moines, Iowa
  - Cotton Oâ€™Neil Diabetes & Endocrinology, Topeka, Kansas
  - Robley Rex VA Medical Center, Louisville, Kentucky
  - MedStar Health Research Institute, Hyattsville, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Profound Research LLC, Clarkston, Michigan
  - Elite Clinical Research Center, Flint, Michigan
  - International Diabetes Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - QCR Network, Omaha, Nebraska
  - Palm Research Center Inc., Las Vegas, Nevada
  - Albuquerque Clinical Trials Inc., Albuquerque, New Mexico
  - AMC Community Endocrinology, Albany, New York
  - NYC Research, Inc., New York, New York
  - NYU Langone Health, New York, New York
  - University at Buffalo, Williamsville, New York
  - Physicians East Endocrinology, Greenville, North Carolina
  - Lucas Research Inc., Morehead City, North Carolina
  - Centricity Res New Bern, New Bern, North Carolina
  - Accellacare Wilmington, Wilmington, North Carolina
  - Diab & Endo Assoc of Stark Co, Canton, Ohio
  - Cleveland Clinic_Cleveland, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Alliance for Multispecialty Research, Norman, Oklahoma
  - Lynn Institute of Norman, Norman, Oklahoma
  - Lynn Institute - East OKC, Oklahoma City, Oklahoma
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Prisma Health Endo Spc Thy Ctr, Greenville, South Carolina
  - Holston Medical Group_Bristol, Bristol, Tennessee
  - University Diabetes & Endocrine Consultants, Chattanooga, Tennessee
  - MidState Endocrine Associates, Nashville, Tennessee
  - Vanderbilt Medical Center_Nashville, Nashville, Tennessee
  - Amarillo Medical Specialists, Amarillo, Texas
  - Texas Diab Endo ATX N Mopac EXPR, Austin, Texas
  - Texas Diabetes & Endocrinology, Austin, Texas
  - Alliance Clinical Network, Dallas, Texas
  - Thyroid Endocrinology & Diabetes PA, Dallas, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Research Institute Of Dallas, Dallas, Texas
  - Precision Endo - Revival, Denton, Texas
  - Epic Medical Research, DeSoto, Texas
  - Frontier Medical Ctr, El Paso, Texas
  - N. Texas Diab & Endo - Prime, Flower Mound, Texas
  - Diabetes and Thyroid Center of Fort Worth, Fort Worth, Texas
  - Houston Endocrinology Center, Houston, Texas
  - The Endocrine Center, Houston, Texas
  - Amir Ali Hassan, MD, PA, Houston, Texas
  - RGV Endocrine Center, McAllen, Texas
  - Tekton Research, McKinney, Texas
  - Be Well Clinical Studies, Round Rock, Texas
  - Texas Diabetes & Endocrinology_Round Rock, Round Rock, Texas
  - Northeast Clinical Research of San Antonio, San Antonio, Texas
  - Valley Diab. & Endo Comp Ctr, Weslaco, Texas
  - Rio Clinical Trials, Ogden, Utah
  - UVM Endocrinology, South Burlington, Vermont
  - Rainier Clin Res Ctr Inc, Renton, Washington
  - Prevea Health, Green Bay, Wisconsin
- Australia (7):
  - Macquarie University, Macquarie Park, New South Wales
  - Illawarra Diabetes Service Clinical Trials & Research Unit, Wollongong, New South Wales
  - Townsville University Hospital, Townsville, Queensland
  - Southern Adelaide Diabetes & Endocrine Services, Oaklands Park, South Australia
  - St Vincent's Hospital - Melbourne, Fitzroy, Victoria
  - Austin Health, Metabolic Disorders Centre, Heidelberg Heights, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- Canada (18):
  - Centricity Research Calgary Endocrinology, Calgary, Alberta
  - University of Calgary, Calgary, Alberta
  - Vancouver General Hospital_Vancouver_0, Vancouver, British Columbia
  - Winnipeg Clinic, Winnipeg, Manitoba
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Centricity Research Brampton Endocrinology, Brampton, Ontario
  - Centricity Research Etobicoke Endocrinology, Etobicoke, Ontario
  - Premier Clinical Trial Research Network (PCTRN), Hamilton, Ontario
  - Western University Centre for Studies in Fam Med, London, Ontario
  - Centricity Research Toronto LMC Multispec, Toronto, Ontario
  - Centricity Research LMC, Toronto, Ontario
  - Ctr de rech Clin de Laval, Laval, Quebec
  - Ctr de recherche Clinique de Laval, Laval, Quebec
  - Centricity Research Mirabel, Mirabel, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Clinique Endocrinologie OASIS., Montreal, Quebec
  - Clin des Mal Lipid de Quebec, Québec, Quebec
  - Centre de Médecine Métabolique de Lanaudière, Terrebonne, Quebec
- Germany (16):
  - Diabetespraxis Mergentheim, Bad Mergentheim
  - Herz- und Diabeteszentrum NRW - Bad Oeynhausen, Bad Oeynhausen
  - Medizinisches Versorgungszentrum Am Bahnhof Spandau GbR, Berlin
  - DSP Bochum, Diabetes- und Stoffwechselpraxis, Bochum
  - Uniklinik TU Dresden - Med. Klinik III, Dresden
  - Praxis für Diabetologie, Angiologie und Innere Medizin Eisenach, Eisenach
  - InnoDiab Forschung GmbH, Essen
  - MVZ Diabeteszentrum Dr. Tews GmbH, Gelnhausen
  - Diabetes-Zentrum-Wilhelmsburg GbR, Hamburg
  - Diabetes Zentrum Wandsbek Berufsausuebungsgemeinschaft GbR, Hamburg
  - Wendisch/Dahl Hamburg (DZHW), Hamburg
  - Die Praxis am Ludwigsplatz, Ludwigshafen
  - MedicalCenter am Clemenshospital - Schwerpunktpraxis für Diabetologie und Ernährungsmedizin, Münster
  - Institut für Diabetesforschung Osnabrück, Osnabrück
  - Zentrum für klinische Studien Alexander Segner, Saint Ingbert-Oberwürzbach
  - Zentrum für klinische Studien Allgäu Oberschwaben, Wangen
- Poland (17):
  - Med. Cent. Diabet. Endo. Metabol. DIAB-ENDO-MET, Krakow, Lesser Poland Voivodeship
  - Formed 2 Sp. z o.o., Oświęcim, Lesser Poland Voivodeship
  - Metabolica Sp. z o.o., Tarnów, Lesser Poland Voivodeship
  - Beata Miklaszewicz & Dariusz Dabrowski "CARDIAMED" s.j., Legnica, Lower Silesian Voivodeship
  - Centrum Medyczne Intercor Sp. z o.o., Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne (UCK), Gdansk
  - Gabinet Lekarski Malgorzata Saryusz-Wolska, Lodz
  - Zanamed Medical Clinic Sp. z o.o., Lublin
  - Reumed Sp. z o.o., Lublin
  - ENDOPRACTICA W.Beker, D.Mielczarek, P.Mielczarek, J.Struzik spolka cywilna, Opole
  - Formed 2 Sp. z o.o., Oświęcim
  - Irmed Klimkiewicz Rudziewicz-Kowalska sp. j., Piotrkow Trybunalski
  - Uniwersyteckie Centrum Stomatologii i Medycyny Specjalistycznej Sp. z o.o., Poznan
  - Gaja Poradnie Lekarskie, Poznan
  - PANSTWOWY INSTYTUT MEDYCZNY MSWiA, Warsaw
  - Zespol Wojewodzkich Przychodni Specjalistycznych W Katowicach SPZOZ, Zabrze
  - Etg Zamosc Sp. z o.o., Zamość
- Puerto Rico (2):
  - Centro de Endo Altagracia, Bayamón
  - Advanced Clinical Research LLC, Bayamón
- Romania (14):
  - S.C. Top Diabet Srl, Craiova, Dolj
  - Diabmed Dr Popescu Alexandrina SRL, Ploieşti, Prahova
  - CMI Dr. Pletea Noemi SRL, Bacau
  - Minimed S.R.L., Bacau
  - Centrul Medical de Diagnostic si Tratament Ambulatoriu Neomed, Brasov
  - SC Nutrilife SRL, Bucharest
  - Diabs&Nutricare Srl, Bucharest
  - Spitalul Clinic Judetean De Urgenta Sfantul Apostol Andrei Constanta, Constanța
  - SC Diamed Obesity SRL, Galati
  - S.C. Dianutrilife Medica S.R.L., Ploieşti
  - Clinica Korall S.R.L. Satu Mare, Satu Mare
  - Spitalul Clinic Judetean de Urgenta Sibiu, Sibiu
  - Spitalul Judetean De Urgenta Sfantul Ioan Cel Nou Suceava, Suceava
  - Spitalul Clinic Judetean De Urgenta Pius Brinzeu Timisoara, Timișoara
- Slovakia (6):
  - DIABEDA s.r.o., Bratislava
  - MEDISPEKTRUM s.r.o., Bratislava
  - Diab - Int, s.r.o., Bytča
  - DIOLI s.r.o., Košice
  - HUMAN-CARE, s.r.o., Košice
  - DIADAN, s.r.o. Kosice, Košice

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com